CLINICAL TRIAL: NCT00323323
Title: A Phase I Study of CHOP and Campath-1H in Previously Untreated Aggressive T/NK-Cell Lymphomas
Brief Title: CHOP and Campath-1H in Previously Untreated Aggressive T/NK-Cell Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0303
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Untreated; CD-20 Negative; Large B-Cell Lymphomas
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Alemtuzumab; Antibodies, Monoclonal, Humanized; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab/CHOP (Experimental): For all patients enrolled, the study will begin with a stepped-up schedule of single agent Alemtuzumab given subcutaneously (SQ) on week #1. Dose escalation will occur during the first week of therapy, starting with 3 mg of Alemtuzumab administered SQ on day 1. If well tolerated, this will be followed by 10 mg SQ on day 3 and 30 mg (split into 2 injection sites) on day 5. Plasma samples will be obtained for Alemtuzumab pharmacokinetics (PK) during the first week of single agent Alemtuzumab stepped up dosing and subsequently before and after the 5th and the 8th Alemtuzumab/CHOP dose
  Interventions: Drug: CHOP; Drug: Alemtuzumab; Procedure: Plasma Samples

INTERVENTIONS:
Drug: CHOP — CHOP will be given 60-120 minutes following SQ administration of Alemtuzumab as follows: cyclophosphamide 750 mg/m2 IV on day 1, doxorubicin 50 mg/m2 IV on day 1, vincristine 1.4 mg/m2 (maximum dose = 2 mg) IV on day 1, and prednisone 100 mg PO on days 1-5.
  Other Names: cyclophosphamide; doxorubicin; vincristine; prednisone
Drug: Alemtuzumab — Single agent Alemtuzumab given subcutaneously (SQ) on week #1. Dose escalation will occur during the first week of therapy, starting with 3 mg of Alemtuzumab administered SQ on day 1. If well tolerated, this will be followed by 10 mg SQ on day 3 and 30 mg (split into 2 injection sites) on day 5.
  Other Names: Humanized monoclonal antibody
Procedure: Plasma Samples — Plasma samples will be obtained for Alemtuzumab pharmacokinetics (PK) during the first week of single agent Alemtuzumab stepped up dosing and subsequently before and after the 5th and the 8th Alemtuzumab/CHOP dose.
  Other Names: Pharmacokinetics; Correlative Studies

SUMMARY:
Purpose: This study will evaluate the safety of CHOP plus Alemtuzumab in patients with T/NK cell lymphomas and CD-20 negative large B-cell lymphomas who have not had previous treatments. The biological response of lymphoma cells and the immune system to this drug combination will also be measured in patients before, during, and after therapy administration.

DETAILED DESCRIPTION:
Rationale: The drug combination called CHOP, or Cyclophosphamide (Cytoxan), Doxorubicin (Adriamycin), Vincristine (Oncovin), and Prednisone (Deltasone), has been used against different types of lymphoma for many years. Researchers are investigating what other therapies to combine with the CHOP regimen to improve outcomes for patients with lymphoma. The current study combines CHOP with alemtuzumab, a monoclonal antibody used against leukemia. Monoclonal antibodies are a type of immunotherapy used against some types of cancer. They are produced in a laboratory and designed to target as well as bind with cells that carry specific proteins. Alemtuzumab is designed to target leukemia cells that express a specific protein. The specific protein recognized by alemtuzumab is the CD52 antigen. This antigen, or substance that causes the immune system to create a specific response, is expressed on normal B and T cells, as well as on abnormal T cells characteristic of certain cancers. Alemtuzumab causes the CD52 antigen to bind with B-cell lymphocytes. This study will also assess the theory that alemtuzumab may increase the effectiveness of the chemotherapy agents included in the CHOP regimen.

Treatment: Patients in this study will receive alemtuzumab and CHOP. Alemtuzumab will be given through injections into the skin and CHOP will be administered through intravenous infusions. Patients will receive alemtuzumab alone during the first week of the study. An increasing amount of alemtuzumab will be given during the first week. If patients cannot tolerate the highest amount of alemtuzumab determined as appropriate within one week, they will be removed from the study. Once the highest dose of alemtuzumab has been achieved, patients will then receive both alemtuzumab and CHOP every three weeks. This schedule will be repeated up to eight times. Several tests and exams will be given throughout the study to closely monitor patients. Treatments will be discontinued due to disease growth or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* CD-20 Negative
* Previous treatment permitted: radiation, electron beam radiotherapy, PUVA, corticosteroids, IFN, low dose methotrexate, retinoids, Ontak
* CNS disease permitted

Exclusion Criteria:

* Pregnant or Nursing
* prior Alemtuzumab
* history of active Hep C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-03; Primary Completion 2012-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Toxicity and safety of concurrent CHOP and Alemtuzumab | up to five years

SECONDARY OUTCOMES:
Determine pharmacokinetics of Alemtuzumab | up to five years
Determine immunosuppressive properties of Alemtuzumab + CHOP | up to five years
Determine if Fc Receptor-gamma (FcγR) polymorphism is predictive of response or toxicity with Alemtuzumab treatment. | up to five years

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Porcu, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu